CLINICAL TRIAL: NCT00235144
Title: E-Sirius Study: a European, Multi-Center, Randomized, Double-Blind Study of the Sirolimus-Coated BX VELOCITY Balloon-Expandable Stent in the Treatment of Patients With de Novo Coronary Artery Lesions
Brief Title: The Study of the BX VELOCITY Stent In Patients With De Novo Coronary Artery Lesions.
Acronym: E-SIRIUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Cordis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC00-07
Record Dates: First submitted 2005-10-04; First posted 2005-10-10 (Estimated); Last update posted 2009-05-11 (Estimated); Status verified 2009-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): drug-eluting stent
  Interventions: Device: sirolimus-coated Bx Velocity stent
- 2 (Active Comparator): bare-metal stent
  Interventions: Device: uncoated Bx Velocity stent

INTERVENTIONS:
Device: sirolimus-coated Bx Velocity stent — drug-eluting stent
  Arms: 1
Device: uncoated Bx Velocity stent — bare-metal stent
  Arms: 2

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the sirolimus-coated Bx VELOCITY™ stent in maintaining minimum lumen diameter in de novo native coronary artery lesions as compared to the uncoated Bx VELOCITY balloon-expandable stent. Both stents are mounted on the Raptor® Rapid Exchange Stent Delivery System.

DETAILED DESCRIPTION:
This is a multicenter (up to 35 centers), prospective, randomized double blind study. This study has a 2-arm design assessing the safety and effectiveness of the sirolimus-coated Bx VELOCITY stent to the uncoated Bx VELOCITY stent, both mounted on the Raptor Rapid Exchange Stent Delivery System. A total of 350 patients will be entered in the study and will be randomized on a 1:1 basis. Patients will be either randomized to the sirolimus coated or uncoated BX-VELOCITY stent. Patients will be followed at 30 days, 6, 9, and 12 months, and at 2, 3, 4, 5, 6, 7, and 8 years post-procedure, with all patients undergoing repeat angiography at 8 months. Medical resource use during the 5 years follow-up period will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II) OR patients with documented silent ischemia;
2. Treatment of a single de novo native coronary artery lesion in a major coronary artery in patients with single or multi-vessel disease; patients with multiple lesions can be included only if the other lesions do not require treatment;
3. Target vessel diameter at the lesion site is >=2.50mm and <=3.0mm in diameter (visual estimate);
4. Target lesion is >=15mm and <=32mm in length (visual estimate);
5. Target lesion stenosis is >50% and <100% (visual estimate);

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK >2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remains above normal at the time of treatment;
2. Has unstable angina classified as Braunwald III B or C and A I-II-III, or is having a peri infarction;
3. Unprotected left main coronary disease with >=50% stenosis;
4. Significant (>50%) stenoses proximal or distal to the target lesion that might require revascularization or impede runoff;
5. Have an ostial target lesion;
6. Angiographic evidence of thrombus within target lesion;
7. Heavily calcified lesion and/or calcified lesion which cannot be successfully predilated;
8. Documented left ventricular ejection fraction <=25%;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2001-03; Primary Completion 2002-10 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
In-stent minimum lumen diameter (MLD). | 8 months.

SECONDARY OUTCOMES:
Composite of MACE defined as death, myocardial infarction (Q wave and non-Q wave), emergent bypass surgery, or repeat TLR. | 1, 6, 9, and 12 months; 2, 3, 4, 5, 6, 7 and 8 years post procedure.
Angiographic binary restenosis (>=50% diameter stenosis). | 8 months.
In-lesion MLD. | 8 months.
Target lesion revascularization. | 9 months.
Target vessel revascularization. | 9 months.
Target vessel failure defined as cardiac death, myocardial infarction, or target vessel revascularization. | 9 months.
Device success (final residual diameter stenosis of < 50%). | any time post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Schofer, MD, Principal Investigator — Herzkatheterlabor und Praxisklinik, Hamburg; Günter Breithardt, MD, Principal Investigator — Med. Klinik und Poliklinik, Münster
Locations (2):
- Germany (2):
  - Herzkatheterlabor und Praxisklinik, Hamburg
  - Med. Klinik und Poliklinik, Münster

REFERENCES:
- [Background] Hoffmann R, Morice MC, Moses JW, Fitzgerald PJ, Mauri L, Breithardt G, Schofer J, Serruys PW, Stoll HP, Leon MB. Impact of late incomplete stent apposition after sirolimus-eluting stent implantation on 4-year clinical events: intravascular ultrasound analysis from the multicentre, randomised, RAVEL, E-SIRIUS and SIRIUS trials. Heart. 2008 Mar;94(3):322-8. doi: 10.1136/hrt.2007.120154. Epub 2007 Aug 29. PMID 17761505
- [Result] Schampaert E, Moses JW, Schofer J, Schluter M, Gershlick AH, Cohen EA, Palisaitis DA, Breithardt G, Donohoe DJ, Wang H, Popma JJ, Kuntz RE, Leon MB; SIRIUS, E- and C-SIRIUS Investigators. Sirolimus-eluting stents at two years: a pooled analysis of SIRIUS, E-SIRIUS, and C-SIRIUS with emphasis on late revascularizations and stent thromboses. Am J Cardiol. 2006 Jul 1;98(1):36-41. doi: 10.1016/j.amjcard.2006.01.049. Epub 2006 May 4. PMID 16784917
- [Result] Schluter M, Schofer J, Gershlick AH, Schampaert E, Wijns W, Breithardt G; E- and C-SIRIUS Investigators. Direct stenting of native de novo coronary artery lesions with the sirolimus-eluting stent: a post hoc subanalysis of the pooled E- and C-SIRIUS trials. J Am Coll Cardiol. 2005 Jan 4;45(1):10-3. doi: 10.1016/j.jacc.2004.09.046. PMID 15629365
- [Result] Schofer J, Schluter M, Gershlick AH, Wijns W, Garcia E, Schampaert E, Breithardt G; E-SIRIUS Investigators. Sirolimus-eluting stents for treatment of patients with long atherosclerotic lesions in small coronary arteries: double-blind, randomised controlled trial (E-SIRIUS). Lancet. 2003 Oct 4;362(9390):1093-9. doi: 10.1016/S0140-6736(03)14462-5. PMID 14550694
- [Derived] Spaulding C, Daemen J, Boersma E, Cutlip DE, Serruys PW. A pooled analysis of data comparing sirolimus-eluting stents with bare-metal stents. N Engl J Med. 2007 Mar 8;356(10):989-97. doi: 10.1056/NEJMoa066633. Epub 2007 Feb 12. PMID 17296825